CLINICAL TRIAL: NCT07240337
Title: Retrospective Evaluation of Muscle Selection, Dosage, and Clinical Outcomes in Botulinum Toxin Applications in Hemiplegic Patients
Brief Title: Botulinum Toxin Applications in Hemiplegic Patients
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: istftreah3
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This retrospective study will be conducted by reviewing the medical records of hemiplegic patients who received botulinum toxin treatment between 2017 and 2020 at the Physical Medicine and Rehabilitation outpatient clinic of Istanbul Physical Medicine and Rehabilitation Training and Research Hospital. A total of 35 hemiplegic patients who underwent botulinum toxin injection and had at least two follow-up records (with a 6-month interval) will be included. Sociodemographic and clinical data, stroke-related characteristics, botulinum toxin dosage, injected muscle groups, medications, and comorbidities will be recorded. Functional assessments, including the Functional Independence Measure (FIM) and Brunnstrom stage, as well as spasticity evaluations using the Modified Ashworth Scale and the Global Spasticity Index, will be obtained from patient files.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years, clinically diagnosed with hemiplegia
* Received botulinum toxin injection for upper and/or lower extremity spasticity
* Availability of recorded data for two time points, including the Functional Independence Measure (FIM), Brunnstrom stage, Modified Ashworth Scale (MAS), Global Spasticity Index (GSI)
* Documentation of injected muscles and total administered botulinum toxin dosage

Exclusion Criteria:

* Missing essential data (e.g., absence of FIM, MAS, GSI, or GAS at either visit)
* Major interventions during the follow-up period such as surgery or initiation of intrathecal baclofen pump therapy
* Severe concomitant neurological disorders (e.g., progressive neurodegenerative diseases) that interfere with assessment

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of hemiplegic patients aged 18-75 years who received botulinum toxin treatment for upper and/or lower extremity spasticity.
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Change in Spasticity Severity: | Baseline
  Evaluated using the Modified Ashworth Scale (MAS) before and after botulinum toxin treatment. A decrease in MAS scores indicates a reduction in muscle tone and improved spasticity control.

SECONDARY OUTCOMES:
Global Spasticity Index (GSI): | Baseline
  Changes in the GSI values before and after treatment will be analyzed to assess overall spasticity reduction.
Functional Independence Measure (FIM): | Baseline
  Functional outcomes will be assessed using FIM scores. An increase in total FIM score indicates improved functional independence.
Brunnstrom Stage: | Baseline
  Motor recovery stages will be evaluated according to the Brunnstrom classification, with higher stages reflecting greater motor improvement.
Injected Muscle Groups and Dosage: | Baseline
  The relationship between injected muscles, total botulinum toxin dosage, and clinical response will be analyzed to identify patterns associated with greater therapeutic benefit.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Physical Medicine and Rehabilitation Research and Training Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)